CLINICAL TRIAL: NCT01775995
Title: Randomized Controlled Trial of Mindfulness Meditation and Cognitive Behavioral Therapy Intervention for Opioid-treated Chronic Low Back Pain
Brief Title: Meditation-CBT for Opioid-treated Chronic Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0656
Record Dates: First submitted 2013-01-22; First posted 2013-01-25 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Pain; Low Back Pain
Keywords: Chronic Pain; Low Back Pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain | interventions — Mindfulness; Meditation; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meditation-CBT (Experimental): Participants receiving the meditation-CBT intervention, in addition to usual care for CLBP and opioid therapy management.
  Interventions: Behavioral: Meditation-CBT Intervention + Usual Care
- Wait-list Control (Other): Participants receiving usual care for CLBP and opioid therapy management.
  Interventions: Other: Usual Care Alone

INTERVENTIONS:
Behavioral: Meditation-CBT Intervention + Usual Care — The intervention combines meditation and standard-of-care CBT strategies for chronic low back pain. It consists of eight weekly 2-hour group sessions guided by trained instructors. In addition to session attendance, experimental participants are asked to practice meditation at home at least 6 days/week, 30 minutes/day during the 26-week study.
  Control participants will be offered the intervention after completing the study.
  All participants receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
  Other Names: Mindfulness Meditation; Meditation; Mindfulness; Usual care; Cognitive Behavioral Therapy
  Arms: Meditation-CBT
Other: Usual Care Alone — All participants receive usual care for opioid-treated CLBP through their regular clinicians, per their recommendations.
  Arms: Wait-list Control

SUMMARY:
Chronic low back pain (CLBP) is one of the most common, costly and disabling conditions. It is often refractory to treatment, with patients requiring long-term opioid therapy. Mindfulness meditation is a promising treatment for chronic pain, mental health and addictive disorders. When combined with cognitive behavioral therapy (CBT), a standard of care for CLBP, it may produce additive benefits. The goal of this randomized controlled trial (RCT) is to evaluate the feasibility and efficacy of an innovative behavioral intervention to improve the health of adults with opioid-treated CLBP. This RCT will test the hypotheses that, at 26 weeks, meditation-CBT group participants (meditation-CBT + usual care), compared to those in a wait-list control group (usual care alone), will improve health-related quality of life (primary outcomes: pain severity and physical function) and reduce opioid medication use (secondary outcome). In addition, they will also decrease alcohol and drug use/misuse, and improve stress-sensitive measures and economic outcomes.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most common, costly and disabling conditions. Treatment for refractory CLBP includes long-term opioid therapy even though it is often only marginally effective. Prescription opioid abuse is a national epidemic. Development of safe, effective non-addictive therapies for chronic pain is a national priority. Mindfulness meditation is a promising, safe treatment for chronic pain, mental health and addictive disorders. When combined with cognitive behavioral therapy (CBT), a standard of care for CLBP, it may produce additive benefits. No study has evaluated the potential of a combined meditation-CBT intervention to improve outcomes in patients with opioid-treated CLBP.

This unblinded 26-week pilot randomized controlled trial (RCT) will test methods feasibility and efficacy of meditation-CBT for improving health-related quality of life (primary outcomes: pain severity and physical function) and reduce opioid medication use (secondary outcome) among adults with opioid-treated CLBP. Eligible participants are adults at least 21 years old, with daily CLBP treated with daily opioids (at least 30 morphine-equivalent mg/day) for at least 3 months. They will be recruited from outpatient clinic and community settings, and randomly assigned to one of two study arms: meditation-CBT + usual care or usual care alone. The targeted meditation-CBT intervention will consist of a) therapist-led group training (two-hours/week for 8 weeks), and b) at-home meditation practice (at least 30 minutes/day, 6 days/week). Control participants will be offered the intervention after their study completion.

Outcome measures, collected at 0, 8 (directly post-intervention) and 26 (18 weeks post-intervention) weeks will gather data on efficacy and potential mechanisms of action of meditation-CBT intervention. This RCT will test the hypotheses that, at 26 weeks, meditation-CBT group participants (meditation-CBT + usual care), compared to those in a wait-list control group (usual care alone), will improve health-related quality of life (primary outcomes: pain severity and physical function) and reduce opioid medication use (secondary outcome). In addition, they will also decrease alcohol and drug use/misuse, and improve stress-sensitive measures and economic outcomes. Increased pain acceptance, mindfulness level or stress reduction are hypothesized to be the mechanistic pathways.

This study directly addresses national priorities aimed at the development of an effective, safe treatment for CLBP and reduction of opioid use. Potential benefits accruing from positive findings include improved quality of life and reduced opioid pain medication use among patients with refractory, opioid-treated CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years old
* Chronic low back pain defined as a daily pain in the lumbosacral region or radiating to the leg (sciatica)
* Pain lasting for and treated with clinician-prescribed daily opioids (≥ 30mg of morphine equivalent dose, MED) for ≥ 3 months
* Has the ability to feel warm and cold temperature sensations in both hands (for pain psychophysical testing)
* English fluent

Exclusion Criteria:

* Experience in meditation (current, regular practice in the past 12 months or past formal training)
* Inability to reliably participate
* Self-reported current pregnancy
* Preexisting delusional, bipolar, or borderline personality disorders
* Individuals lacking consent capacity and prisoners

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Zgierska, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Background] Dr. Zgierska was supported by the K23AA017508 from the National Institutes of Health (NIH) National Institute on Alcohol Abuse and Alcoholism (NIAAA). The project was also supported by the Clinical and Translational Science Award (CTSA) program through the NIH National Center for Advancing Translational Sciences (NCATS), grant UL1TR000427. The content is solely the responsibility of the authors and does not necessarily represent the official views of the NIH.
- [Derived] Zgierska AE, Burzinski CA, Cox J, Kloke J, Stegner A, Cook DB, Singles J, Mirgain S, Coe CL, Backonja M. Mindfulness Meditation and Cognitive Behavioral Therapy Intervention Reduces Pain Severity and Sensitivity in Opioid-Treated Chronic Low Back Pain: Pilot Findings from a Randomized Controlled Trial. Pain Med. 2016 Oct;17(10):1865-1881. doi: 10.1093/pm/pnw006. Epub 2016 Mar 10. PMID 26968850

RESULTS

PARTICIPANT FLOW:
Groups:
- Meditation-CBT: Meditation-CBT + Usual Care
  Participants receiving the meditation-CBT intervention, in addition to usual care for CLBP and opioid therapy management.
- Wait-list Control: Usual Care
  Participants receiving usual care for CLBP and opioid therapy management.
Period: Overall Study
Arm/Group | Meditation-CBT | Wait-list Control
Started | 21 | 14
Completed | 20 (One experimental participant was unable to reach at 26 week follow up) | 13 (One control participant was unable to reach at 26 week follow up)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Meditation-CBT: Mindfulness-CBT + Standard of Care Therapy
  Mindfulness Based Intervention with Cognitive Behavioral Therapy (CBT) components: All study subjects receive standard of care therapy. In addition, experimental subjects receive the mindfulness-CBT. The intervention consists of an 8-week meditation-CBT course (2 hour weekly group sessions) and daily, at-home practice (30 mins/day, 6 days/week of formal practice). Controls will be offered meditation intervention after completing the study.
- Wait-list Control: Standard of Care Therapy only
- Total: Total of all reporting groups
Arm/Group | Experimental: Meditation-CBT | Wait-list Control | Total
Number analyzed (Participants) | 21 | 14 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.5) | 50.5 (8.6) | 51.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 13 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 16 | 12 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 14 | 35
Physical Function [Mean (Standard Deviation); unit: percent] — Physical function was assessed using the 10-item Oswestry Disability Index. This measure's total score (0-100) reflects the percent of chronic low back pain related disability "today". Zero to 20% is considered "minimal disability", 21 to 40% "moderate disability", 41 to 60% "severe disability", 61 to 80% "crippled", and 81 to 100% "bed bound".
  percent | 68.1 (9.3) | 64.5 (14.1) | 66.7 (11.4)
Averaged Pain [Mean (Standard Deviation); unit: units on a scale] — Averaged pain is the average of 4 responses on a 0-10 numerical rating scale (0=no pain; 10=worst possible pain) from the Brief Pain Inventory (BPI): 1) describe your pain at its worst in the last week 2) describe your pain at its least in the last week 3) describe your pain on the average 4) describe your pain right now.
  units on a scale | 6.3 (1.2) | 4.9 (1.1) | 5.8 (1.4)
Opioid Use [Mean (Standard Deviation); unit: mg/day] — Opioid use was measured using the Timeline Followback Method which looked at the past 28 days of opioid use. Opioid use was standardized [daily morphine-equivalent dose (MED)] across different opioids for each participant.
  mg/day | 166.9 (153.7) | 120.3 (76.9) | 148.3 (129.2)

OUTCOME MEASURES:

1. Primary Outcome: Health-Related Quality of Life: Averaged Pain Severity
Description: Averaged pain is the average of 4 responses on a 0-10 numerical rating scale (0=no pain; 10=worst possible pain) from the Brief Pain Inventory (BPI): 1) describe your pain at its worst in the last week 2) describe your pain at its least in the last week 3) describe your pain on the average 4) describe your pain right now.
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased pain and negative values indicating decreased pain.
Time Frame: baseline to 8 weeks
Population: One Meditation-CBT participant did not provide data for this measure at 8-week follow up. Results on this measure are based on the number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | -0.5 [-1.1 to 0.03] | 0.4 [-0.3 to 1.0]

2. Primary Outcome: Health-Related Quality of Life: Averaged Pain Severity
Description: Averaged pain is the average of 4 responses on a 0-10 numerical rating scale (0=no pain; 10=worst possible pain) from the Brief Pain Inventory (BPI): 1) describe your pain at its worst in the last week 2) describe your pain at its least in the last week 3) describe your pain on the average 4) describe your pain right now.
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased pain and negative values indicating decreased pain.
Time Frame: baseline to 26 weeks
Population: One Meditation-CBT and one Wait-list Control participant did not provide data for this measure at 26-week follow up. Results on this measure are based on the number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -0.5 [-1.1 to 0.02] | 0.5 [-0.2 to 1.2]

3. Primary Outcome: Health-Related Quality of Life: Physical Function
Description: Physical function was assessed using the 10-item Oswestry Disability Index (ODI). This measure's total score (0-100) reflects the percent of chronic low back pain related disability "today".
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased disability and negative values indicating decreased disability.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage disability
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
percentage disability | -2.4 [-7.2 to 2.3] | -0.6 [-6.2 to 5.1]

4. Primary Outcome: Health-Related Quality of Life: Physical Function
Description: Physical function was assessed using the 10-item Oswestry Disability Index (ODI). This measure's total score (0-100) reflects the percent of chronic low back pain related disability "today".
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased disability and negative values indicating decreased disability.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage disability
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
percentage disability | -5.0 [-9.7 to -0.2] | 1.6 [-4.3 to 7.4]

5. Secondary Outcome: Opioid Dose
Description: Daily opioid dose was assessed using the Timeline Followback Method which looked at the past 28 days of opioid use. Medication use reports were verified against the medication bottles. Daily opioid dose was standardized [daily morphine-equivalent dose (MED)] across different opioids for each participant.
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased daily opioid dose and negative values indicating decreased daily opioid dose.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: morphine-equivalent mg/day
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
morphine-equivalent mg/day | -7.1 [-32.5 to 18.3] | -1.4 [-32.3 to 29.5]

6. Secondary Outcome: Opioid Dose
Description: Daily opioid dose was assessed using the Timeline Followback Method which looked at the past 28 days of opioid use. Medication use reports were verified against the medication bottles. Daily opioid dose was standardized [daily morphine-equivalent dose (MED)] across different opioids for each participant.
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased daily opioid dose and negative values indicating decreased daily opioid dose.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: morphine-equivalent mg/day
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
morphine-equivalent mg/day | -10.1 [-35.5 to 15.2] | -0.2 [-31.4 to 30.9]

7. Other Pre Specified Outcome: Alcohol Use
Description: Percentage of participants endorsing any alcohol use during the past 28 days was assessed using the Timeline Follow-Back Method.
Time Frame: Baseline
Measure: Number; unit: percentage using alcohol
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 21 | 14
percentage using alcohol | 28.6 | 21.4

8. Other Pre Specified Outcome: Alcohol Use
Description: as for outcome 7
Time Frame: 8 weeks
Population: One Meditation-CBT participant did not provide data for this measure at 8 week follow-up. Results for this measure are based on the number of participants analyzed.
Measure: Number; unit: percentage using alcohol
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
percentage using alcohol | 30.0 | 42.9

9. Other Pre Specified Outcome: Alcohol Use
Description: as for outcome 7
Time Frame: 26 weeks
Population: One Meditation-CBT and one Wait-list Control participant did not provide data for this measure at 26 week follow-up. Results for this measure are based on the number of participants analyzed.
Measure: Number; unit: percentage using alcohol
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
percentage using alcohol | 20.0 | 38.5

10. Other Pre Specified Outcome: Drug Use
Description: Percentage of participants endorsing drug use during the past 28 days was assessed using the Timeline Follow-Back Method.
Time Frame: Baseline
Measure: Number; unit: percentage using drugs
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 21 | 14
percentage using drugs | 28.6 | 14.2

11. Other Pre Specified Outcome: Drug Use
Description: as for outcome 10
Time Frame: 8 weeks
Population: as for outcome 8
Measure: Number; unit: percentage using drugs
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
percentage using drugs | 35.0 | 7.1

12. Other Pre Specified Outcome: Drug Use
Description: as for outcome 10
Time Frame: 26 weeks
Population: as for outcome 9
Measure: Number; unit: percentage using drugs
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
percentage using drugs | 30.0 | 7.7

13. Other Pre Specified Outcome: Chronic Pain Acceptance
Description: Pain acceptance was assessed using the 20-item Chronic Pain Acceptance Questionnaire (CPAQ). This measure's total score (0-120) reflects one's degree of acceptance of their chronic pain, not specifying a time frame.
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased chronic pain acceptance and negative values indicating decreased chronic pain acceptance.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | 5.9 [-0.6 to 12.4] | 3.2 [-4.7 to 11.2]

14. Other Pre Specified Outcome: Chronic Pain Acceptance
Description: Pain acceptance was assessed using the 20-item Chronic Pain Acceptance Questionnaire (CPAQ). This measure's total score (0-120) reflects one's degree of acceptance of their chronic pain, not specifying a time frame.
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased chronic pain acceptance and negative values indicating decreased chronic pain acceptance.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | 14.7 [8.1 to 21.2] | 9.3 [1.3 to 17.4]

15. Other Pre Specified Outcome: Perceived Stress
Description: Perceived stress was assessed using the 10-item Perceived Stress Scale (PSS-10). This measure's total score (0-40) reflects the degree to which one perceives their life experiences as stressful "in the last month".
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased perceived stress and negative values indicating decreased perceived stress.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | 0.6 [-2.5 to 3.6] | 0.2 [-3.5 to 3.9]

16. Other Pre Specified Outcome: Perceived Stress
Description: Perceived stress was assessed using the 10-item Perceived Stress Scale (PSS-10). This measure's total score (0-40) reflects the degree to which one perceives their life experiences as stressful "in the last month".
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased perceived stress and negative values indicating decreased perceived stress.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -1.7 [-4.8 to 1.3] | -1.8 [-5.6 to 2.0]

17. Other Pre Specified Outcome: Mental Health Symptom Severity
Description: Mental Health Symptom Severity was assessed using the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's Global Severity Index (i.e. total score, 0-360) reflects the degree of severity of mental health symptom distress "during the past 7 days".
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased levels of mental health symptom distress and negative values indicating decreased mental health symptom distress.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | -0.03 [-0.2 to 0.1] | -0.1 [-0.3 to 0.1]

18. Other Pre Specified Outcome: Mental Health Symptom Severity
Description: Mental Health Symptom Severity was assessed using the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's Global Severity Index (i.e. total score, 0-360) reflects the degree of severity of mental health symptom distress "during the past 7 days".
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased levels of mental health symptom distress and negative values indicating decreased mental health symptom distress.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -0.2 [-0.3 to -0.01] | -0.3 [-0.5 to -0.04]

19. Other Pre Specified Outcome: Depression Symptom Severity
Description: Depression symptom severity was assessed using the depression subscale of the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's 13-item Depression subscale (0-52) reflects the degree of severity of distress from depression symptoms "during the past 7 days".
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased levels of distress from depression symptoms and negative values indicating decreased levels of distress from depression symptoms.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | 0.04 [-0.2 to 0.3] | -0.1 [-0.5 to 0.2]

20. Other Pre Specified Outcome: Depression Symptom Severity
Description: Depression symptom severity was assessed using the depression subscale of the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's 13-item Depression subscale (0-52) reflects the degree of severity of distress from depression symptoms "during the past 7 days".
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased levels of distress from depression symptoms and negative values indicating decreased levels of distress from depression symptoms.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -0.3 [-0.6 to 0.02] | -0.4 [-0.7 to -0.02]

21. Other Pre Specified Outcome: Anxiety Symptom Severity
Description: Anxiety symptom severity was assessed using the anxiety subscale of the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's 10-item Anxiety subscale (0-40) reflects the degree of severity of distress from anxiety symptoms "during the past 7 days".
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased levels of distress from anxiety symptoms and negative values indicating decreased levels of distress from anxiety symptoms.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | -0.2 [-0.4 to 0.1] | -0.3 [-0.5 to 0.03]

22. Other Pre Specified Outcome: Anxiety Symptom Severity
Description: Anxiety symptom severity was assessed using the anxiety subscale of the 90-item Symptom Checklist - Revised (SCL-90-R). This measure's 10-item Anxiety subscale (0-40) reflects the degree of severity of distress from anxiety symptoms "during the past 7 days".
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased levels of distress from anxiety symptoms and negative values indicating decreased levels of distress from anxiety symptoms.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -0.2 [-0.4 to 0.05] | -0.3 [-0.5 to 0.02]

23. Other Pre Specified Outcome: Emotion Regulation Difficulty
Description: Emotion regulation difficulty was assessed using the 36-item Difficulties in Emotion Regulation Scale (DERS). This measure's total score (36-180) reflects the severity of emotion regulation difficulty (no timeframe specified).
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure), with positive values indicating increased emotion regulation difficulty and negative values indicating decreased emotion regulation difficulty.
Time Frame: baseline to 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 14
units on a scale | -0.8 [-8.3 to 6.7] | -1.6 [-10.7 to 7.5]

24. Other Pre Specified Outcome: Emotion Regulation Difficulty
Description: Emotion regulation difficulty was assessed using the 36-item Difficulties in Emotion Regulation Scale (DERS). This measure's total score (36-180) reflects the severity of emotion regulation difficulty (no timeframe specified).
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure), with positive values indicating increased emotion regulation difficulty and negative values indicating decreased emotion regulation difficulty.
Time Frame: baseline to 26 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 20 | 13
units on a scale | -4.0 [-11.7 to 3.6] | -4.2 [-13.5 to 5.1]

25. Other Pre Specified Outcome: C-Reactive Protein
Description: Serum levels of C-reactive protein were used to assess the potential biological effects of the intervention. Normal values for C-reactive protein fall between 0 and 1 mg/dL; higher levels may indicate inflammatory or infectious processes.
  This outcome measure for 8 week follow up is expressed as a difference score (change from baseline to 8 week measure).
Time Frame: baseline to 8 weeks
Population: Three Meditation-CBT participants did not provide biological data at 8 week follow-up. Results for this measure are based on the number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 18 | 14
mg/dL | -0.9 [-1.7 to -0.1] | 0.1 [-0.9 to 1.0]

26. Other Pre Specified Outcome: C-Reactive Protein
Description: Serum levels of C-reactive protein were used to assess the potential biological effects of the intervention. Normal values for C-reactive protein fall between 0 and 1 mg/dL; higher levels may indicate inflammatory or infectious processes.
  This outcome measure for 26 week follow up is expressed as a difference score (change from baseline to 26 week measure).
Time Frame: baseline to 26 weeks
Population: Six Meditation-CBT participants and one Wait-list Control participant did not provide biological data at 26 week follow-up. Results for this measure are based on the number of participants analyzed.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 15 | 13
mg/dL | -0.7 [-1.6 to 0.1] | 0.1 [-0.9 to 1.0]

27. Other Pre Specified Outcome: Economic Outcomes
Description: Cost of medications, health care utilization, motor vehicle accidents (MVAs), and lost productivity were assessed.
  Medications (past month - self-report, verified against medication bottles): opioids (Timeline Followback), other medications (average daily use); costs for the past 6 months were calculated. Health care utilization (past 6 months): self-reported number of outpatient (medical, mental health, urgent care) and emergency department visits; number of inpatient days. Lost productivity (past 6 months): self-report number of missed work and leisure days. MVAs (past 6 months): self-report number of MVAs.
  Cost Sources: Medications - rxpricequotes.com (primary), drugs.com (secondary), walgreens.com (tertiary). Health care utilization - WI Price Point System, Medical Expenditure Panel Survey. MVAs - National Safety Council. Lost productivity - U.S. Dept of Labor (average daily wage for a WI worker for work days; 8-hours of the federal minimum wage for lost leisure day).
Time Frame: 6 months prior to baseline, to baseline (enrollment)
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 21 | 14
dollars | 16443 (15634) | 14284 (11091)

28. Other Pre Specified Outcome: Economic Outcomes
Description: as for outcome 27
Time Frame: From enrollment to 26 week follow-up (6 months)
Population: One meditation-CBT participant did not provide data at 8-week follow-up; two participants (one meditation-CBT, one control) did not provide data at 26-week follow-up. All 35 participants were included in the analysis; missing participant data was imputed based on existing data for the given participant.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Meditation-CBT | Wait-list Control
Number analyzed (Participants) | 21 | 14
dollars | 11576 (8347) | 11697 (9876)

29. Other Pre Specified Outcome: Pain Sensitivity to Experimental Thermal Stimuli
Description: Pain sensitivity to thermal stimuli was assessed using standard psychophysical procedures. Thermal stimuli, ranging from 43 to 49oC, were applied to the thenar eminence of the right hand. Each stimulus was rated on two separate, validated 0-20 category-ratio scales assessing pain intensity and unpleasantness.
Time Frame: 0, 8, 26 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Experimental: Meditation-CBT | Wait-list Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 7/21 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Meditation-CBT (N=21) | Wait-list Control (N=14)
Increased cigarette smoking (General disorders) | 1 (1) | 0 (0) — One participant reported increased cigarette smoking during the meditation course (course started on 3-25-13), however, prior to the end of the course this individual reported they were able to quit smoking altogether (on 5-1-13).
Weight gain (General disorders) | 1 (1) | 0 (0) — One participant reported an increase in weight during the meditation course (course started on 3-25-13), however after the end of the course the participant reported their weight decreased again (on 5-21-13).
Increased pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Two participants reported increased pain with mindful movement or when learning to mindfully 'observe' pain experiences, during the meditation course (course started on 3-25-13 and ended on 5-13-13).
Anxiety/Emotional Distress (General disorders) | 3 (3) | 0 (0) — Three participants reported increased anxiety or emotional distress while learning the meditation intervention techniques during the course (course started on 3-25-13 and ended on 5-13-13).

LIMITATIONS AND CAVEATS:
Lack of blinding of study staff to group status (except the statistician who was blinded during initial primary analyses); conducting most study related activities by the same core group of research staff may have introduced bias and placebo effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes